CLINICAL TRIAL: NCT02521688
Title: Inflammatory Cytokines in Gingival Crevicular Fluid and Placental Tissues in Chronic Periodontitis Patients With Preterm Delivery
Brief Title: Inflammatory Cytokines in GCF and Placental Tissues in Chronic Periodontitis Patients With Preterm Delivery
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ola Mohamed Ezzatt, lecturer of oral medicine and periodontology, Ain Shams University
Other Study IDs: FDASU-RECD 1214402
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Preterm Labor; Periodontitis
MeSH Terms: conditions — Obstetric Labor, Premature; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Placental tissue Gingival clevicular fluid from deepest pocket
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I (PTD + CP): include ten mothers exhibiting spontaneous preterm delivery with moderate to severe chronic periodontitis +incisional biopsy from placenta and GCF sample
  Interventions: Procedure: incisional biopsy from placenta and GCF sample
- Group II (TD + CP): include ten mothers exhibiting spontaneous term delivery with moderate to severe chronic periodontitis+incisional biopsy from placenta and GCF sample
  Interventions: Procedure: incisional biopsy from placenta and GCF sample
- Group III (PTD + HP): include tenmothersexhibiting spontaneous preterm delivery with healthy periodontium +incisional biopsy from placenta and GCF sample
  Interventions: Procedure: incisional biopsy from placenta and GCF sample
- Group IV (TD + HP): ten mothersexhibiting spontaneous term delivery with healthy periodontium(Armitage GC. 1999)+ incisional biopsy from placenta and GCF sample
  Interventions: Procedure: incisional biopsy from placenta and GCF sample

INTERVENTIONS:
Procedure: incisional biopsy from placenta and GCF sample — A small piece of villous placental tissue (approximately 1 cm3) will be dissected free of maternal decidua from the placental bed after delivery of fetus processed to prepare tissue homogenate according to the standardized technique (Keelan JA, et al. 1999) GCF will be obtained from each patient by filter paper inserted in gingival crevice for few seconds after isolation by cotton.

SUMMARY:
Investigators have shown the presence of elevated proinflammatory cytokines in amniotic fluid in patients in preterm labor.However, there is limited and mostly negative evidence that the elevation of these mediators in gingival crevicular fluid (GCF), and amniotic fluid are associated with pregnancy complications in periodontitis patients. Thus this case control study will be conducted to

1. To determine the level of proinflammatory cytokines in gingival crevicular fluid in women with spontaneous preterm delivery with chronic periodontitis.
2. To investigate the expression of macrophage inflammatory protein-1α in placental tissues.
3. To assess the possible correlation between chronic periodontitis and preterm delivery.

DETAILED DESCRIPTION:
Periodontal disease is a commonGram-negative chronic anaerobic infection of the periodontium, with an estimatedworld prevalence of 10% to 15% (Genco RJ, et al. 1992, Petersen PE & Ogawa H. 2005). It Involves both direct tissue damage resulting from plaque bacterial products, and indirect damage via host inﬂammatory and immune responsesmediated by interactions between numerous cell populations and inflammatory mediators (Yucel-Lindberg T&Båge T.2013).

Periodontal infections have been associated with different systemic diseases; cardiovascular disease, cerebrovascular disease, diabetes mellitus, respiratory infections and others including osteoporosis, cancer, rheumatoid arthritis, erectile dysfunction, Alzheimer's disease, gastrointestinal disease, prostatitis and renal diseases(Gulati M, et al. 2013). Moreover, many investigators have reported an association between periodontal disease and adverse pregnancy outcomes, including preterm birth, low birth weight, foetal growth restriction, preeclampsia and perinatal mortality (Ide M&Papapanou PN.2013).

Preterm birth, defined as a live birth before 37 weeks of gestation, is the leading cause of infant mortality in both developed and developing countries (Saigal S & Doyle LW. 2008), whether following spontaneous preterm labour, premature rupture of membranes, or caesarean section due to foetal distress or maternal medical conditions (Goldenberg RL, et al. 2008).The World Health Organization has recently estimated that annually 12.9 million or 9.6% of all children are born preterm worldwide, despite extensive research and public health efforts(Beck S, et al. 2010).

Major causes for preterm birth are intra-amniotic infections which subsequently cause inflammation, as well as sterile inflammation (Madan I, et al 2010). Moreover, smoking, alcohol consumption, black race, low socio-economic status, low or high maternal body mass index, stress, previous preterm birth, advanced maternal age and short cervix are other associated risk factors (DjelantikA, et al. 2012).

Offenbacher et al in 1996 first hypothesized that gram-negative anaerobic pathogens from periodontium and associated endotoxins and maternal inflammatory mediators could have a possible adverse effect on the developing fetus (Offenbacher S, et al. 1996), whether through translocation of periodontal pathogens to the feto-placental unit or the action of the periodontal reservoir of inﬂammatory mediators, which elaborated at the remote site of infection and trigger prostaglandins synthesis, resulting in cervical dilation, entry of more microbes into the uterus, and continuation of the "viscous cycle" resulting in premature birth (Gibbas RS, 2001).

Investigators have shown the presence of elevated proinflammatory cytokines in amniotic fluid, such as interleukin-1α (IL-1α), interleukin-1β (IL-1β), interleukin-6 (IL-6), interleukin-8 (IL-8), and tumor necrosis factor alpha (TNF-α) in patients in preterm labor(Hillier SL, et al. 1993, Hitti J, et al. 2001, Figueroa R, et al. 2005).However, there is limited and mostly negative evidence that the elevation of these mediators in gingival crevicular fluid (GCF), and amniotic fluid are associated with pregnancy complications in periodontitis patients(Madianos PN, et al. 2013).

Macrophage inflammatory proteins 1 alpha (MIP-1α/CCL3) is a member of the cysteine-cysteine chemokine family which is secreted by macrophages, neutrophils, basophils, dendritic cells, lymphocytes and epithelial cells and mediates granulocyte migration and adhesion. It stimulates monocytes and/or osteoclast progenitor cells to become active osteoclasts(Menten P, et al. 2002), as well as regulating hematopoiesis and stimulating production of other inflammatory mediators such as IL-1, TNF alpha(Maurer M & von Stebut E. 2004).

The Level of MIP-1 in GCF found to discriminate between diseased and healthy periodontal sites(Tymkiw KD, et al. 2011). Moreover, its presence whether in cord blood or amniotic fluid was elevated in cases of preterm labor (Matoba N, et al 2009, Weissenbacher T, et al. 2013).

Deliveries prior to 35 weeks of gestation was typically associated with subclinical chorioamnionitis, which is considered the most common manifestation and is defined histologically by inflammation of the chorion, amnion, and placenta, and found to be associated with chronic infections of low virulence organisms (Hagberg H, et al. 2002). However, variability in the assessment criteria for the diagnosis of histological chorioamnionitis exists within the literature (Holzman C, et al. 2007).

Since 1996, a number of studies have investigated the potential relationship between periodontitis and preterm and low birth weight. However, results have been controversial, suggesting the need for more research to confirm or discard this association(Sanz M, et al 2013). Thus this case control study will be conducted to investigate the association between chronic periodontitis and preterm labor through possible correlation between Macrophage Inflammatory Protein-1 alpha (MIP-1α), Tumor necrosis factor alpha (TNF-α) and pentrixin 3 in placental tissues and its level in GCF.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing spontaneous term delivery (TD) at ≥37 weeks of gestation without any obstetrical or medical complications or spontaneous preterm delivery (PTD)at< 37 weeks of gestation after uterine contraction or rupture of membranes(Keelan JA, et al. 1999).
* With a body mass index (BMI) ranged from 19-25.
* Having no systemic disease as evidenced by Burkett's oral medicine health history questionnaire (Glick et al, 2008).

Exclusion Criteria:

* Mothers receiving antibiotics or corticosteroids during last three months of pregnancy or at delivery.
* Current Smokers and drug abusers or stopped from period shorter than 6 months.
* Mothers with urinary tract infection, vulvovaginal infection, previous preterm birth, or any othermedical disorder associated with pregnancy as obtained from patient's record.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fourty Mothers participating in this study recruited from Maternal-Fetal medicine clinic, Faculty of Medicine, Ain Shams University that must undergo delivery without induction, i.e. delivery following labour pains not pre-scheduled caesarian sections
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proinflammatory cytokine level | 1 year
  MIP, TNF, Pentrixin 3 measured in placental tissue homogenate and in GCF